CLINICAL TRIAL: NCT00099970
Title: Phase II Open-Label Study of Volociximab in Combination With DTIC in Patients With Metastatic Melanoma Not Previously Treated With Chemo
Brief Title: Volociximab in Combination With DTIC in Patients With Metastatic Melanoma Not Previously Treated With Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PDL BioPharma, Inc. (Industry)
Organization: Facet Biotech (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M200-1203
Record Dates: First submitted 2004-12-21; First posted 2004-12-22 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Melanoma; Metastases
Keywords: Solid tumors; Metastatic melanoma
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — volociximab; Dacarbazine

INTERVENTIONS:
Drug: M200 (volociximab) in Combination with Dacarbazine (DTIC)

SUMMARY:
This clinical trial is being conducted to determine tumor response and preliminary safety of a monoclonal antibody that specifically binds to a cell surface receptor (α5β1 integrin) that is required for the establishment of new blood vessels during tumor growth, a process known as angiogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of at least 18 years of age with stage IV or unresectable stage III non-ocular melanoma who may have received 0 to 2 prior regimens for metastatic disease with a biological therapy or immunotherapy (e.g., IL-2 or interferon-alfa).
* Measurable disease according to Response Criteria for Solid Tumors (RECIST).
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1.
* Estimated survival is greater or equal to 4 months.
* Negative pregnancy test (women of childbearing potential only).
* Pretreatment laboratory levels that meet specific criteria.
* Signed informed consent, including permission to use protected health information.

Exclusion Criteria:

* Prior treatment with M200 or a5b1 inhibitors and murine or chimeric monoclonal antibodies.
* Prior treatment with DTIC, temozolomide, or other chemotherapeutic regimens.
* Known sensitivity to murine proteins or chimeric antibodies or other components of the product.
* Use of any investigational drug within 4 weeks prior to screening or 5 half-lives of the prior investigational drug (whichever is longer).
* Systemic biologic, immunotherapy, and/or radiation therapy within 4 weeks of the first dose of M200.
* Documented central nervous system (CNS) tumor or CNS metastasis.
* History of thromboembolic events and bleeding disorders within the past year.
* Medical conditions that may be exacerbated by bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-12; Study Completion 2006-03

PRIMARY OUTCOMES:
Proportion of patients with a confirmed tumor response at any time during the study.

SECONDARY OUTCOMES:
Time to disease progression
Duration of tumor response
Pharmacokinetics (PK)
Immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Steven J. O'Day, M.D., Principal Investigator — Cancer Institute Medical Group, Inc.; John Kirkwood, M.D., Principal Investigator — University of Pittsburgh; Agop Y. Bedikian, MD, Principal Investigator — M.D. Anderson Cancer Center; Antoni Ribas, MD, Principal Investigator — University of California, Los Angeles; Colin P. Curran, M.D., Principal Investigator — Palmetto Hematology Oncology, P.C.; Andres Forero, M.D., Principal Investigator — University of Alabama at Birmingham; Lee Cranmer, M.D., Principal Investigator — University of Arizona
Locations (7):
- United States (7):
  - University of Alabama at Birmingham-Comprehensive Cancer Ctr., Birmingham, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - UCLA School of Medicine, Los Angeles, California
  - Cancer Institute Medical Group, Inc., Santa Monica, California
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Palmetto Hematology Oncology, P.C., Spartanburg, South Carolina
  - MD Anderson Cancer Center, Houston, Texas